CLINICAL TRIAL: NCT06163196
Title: The Effect Of Acupressure Application On Reducing Pain During Venipuncture İn Children Dıagnosed With Thalassemia.
Brief Title: The Effect of Acupressure on Pain in Children With Thalassemia
Acronym: acupressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Melek Gulgun Altintas, Principal investigator, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: j94ghcf2
Record Dates: First submitted 2022-12-11; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Pain
Keywords: acupressure; thalassemia; child; pediatric nursing
MeSH Terms: conditions — Pain; Thalassemia | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: prospective, parallel , randomized controlled clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Since there are 40 children with a diagnosis of Thalassemia in total, aged between 6-18 years, who applied to Mersin City Training and Research Hospital Pediatric Hematology Polyclinic and Daily Pediatric Service between 7 February and 4 June 2022, agreed to participate in the study, and gave permission from their parents, without sampling. 39 children participated. The acupressure group consisted of 19 children and the placebo group consisted of 20 children. During the procedure, children were taken into the room where blood collection took place, one by one, together with their parents. Thus, children and parents participating in the study were prevented from influencing each other. During the application and analysis processes of the research, the groups represented by the papers written "Group A" and "Group B" were blinded and hidden from the child who agreed to participate in the research, the parents, and the statistician who performed the analyses.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- accupressure (Experimental): In the study group (n:19), blood pressure, pulse and oxygen saturation were measured, and the acupressure points determined (large intestine meridian 4. Point: LI 4, large intestine meridian 11. Point: LI 11, Heart Meridian 7. Point: HT 7 ) acupressure was applied for only one session by applying light pressure with the thumb of the practitioner's hand, in two directions as the right and left arms, for 2 minutes to each point for a total of 12 minutes. Blood was drawn immediately after the procedure. In order to evaluate the child's pain immediately after the blood collection procedure, the child was asked to mark the most appropriate face on the Wong Baker Faces Pain Rating Scale. In addition, the child's pain was evaluated by the researcher and the parent using the Wong Baker Faces Pain Rating Scale. After the pain assessment, the child's heart rate, oxygen saturation and blood pressure were re-evaluated by the researcher and recorded in the Procedure Record Form.
  Interventions: Other: acupressure
- control (Sham Comparator): The point used in our research is the point located in the middle of the third and fourth metacarpal bones on the back of the hand. Children in the placebo control group (n:20) were touched by the researcher for one minute without applying pressure or massage to the determined placebo point immediately after their physiological parameters were evaluated. Immediately after blood collection, the child was asked to mark the most appropriate facial expression on the Wong Baker Faces Pain Rating Scale so that he or she could assess his pain. In addition, the child's pain was evaluated by the researcher and the parent using the Wong Baker Faces Pain Rating Scale.
  Interventions: Other: acupressure

INTERVENTIONS:
Other: acupressure — Before the blood collection procedure, pressure will be applied to the acupressure points determined by the researcher for 2 minutes and then blood collection will be performed.

SUMMARY:
This randomized controlled trial evaluates the effect of acupressure on reducing the pain of blood collection in children with Thalassemia. The hypothesis of this study is that acupressure application reduces acute pain.

DETAILED DESCRIPTION:
A total of 39 children with a diagnosis of Thalassemia were randomly assigned to the study and control groups. In the study group (n:19), blood pressure, pulse and oxygen saturation were measured, and the acupressure points determined (large intestine meridian 4. Point: LI 4, large intestine meridian 11. Point: LI 11, Heart Meridian 7. Point: HT 7 ) acupressure was applied for only one session by applying light pressure with the thumb of the practitioner's hand, in two directions as the right and left arms, for 2 minutes to each point for a total of 12 minutes. Blood was drawn immediately after the procedure. In order to evaluate the child's pain immediately after the blood collection procedure, the child was asked to mark the most appropriate face on the Wong Baker Faces Pain Rating Scale. In addition, the child's pain was evaluated by the researcher and the parent using the Wong Baker Faces Pain Rating Scale. After the pain assessment, the child's heart rate, oxygen saturation and blood pressure were re-evaluated by the researcher and recorded in the Procedure Record Form.

Placebo (sham) acupressure application is the pressure of the fingers on the non-meridian region without a specific acupressure point. The point used in our research is the point located in the middle of the third and fourth metacarpal bones on the back of the hand. The children in the placebo control group were only touched by the researcher without applying pressure and massage for one minute to the determined placebo point immediately after their physiological parameters were evaluated, and immediately after that, blood collection was performed. Immediately after blood collection, the child was asked to mark the most appropriate facial expression on the Wong Baker Faces Pain Rating Scale so that he or she could evaluate his pain. In addition, the child's pain was evaluated by the researcher and the parent using the Wong Baker Faces Pain Rating Scale. After the pain assessment, the child's heart rate, oxygen saturation and blood pressure were re-evaluated by the researcher and recorded in the Procedure Record Form.

ELIGIBILITY:
Inclusion Criteria:

* Registered in the centers where the study will be carried out,
* Able to communicate verbally
* No developmental or sensory disabilities,
* No mental illness
* No opioid, narcotic analgesic or sedative use in the last 8 hours before the procedure,
* No other chronic disease
* One-time bloodletting
* Children who agree to participate in the study.

Exclusion Criteria:

* Having pain before the blood draw procedure,
* Not between the ages of 6-18,
* Have developmental or sensory disabilities,
* Having a mental illness
* Using opioids, narcotic analgesics or sedatives in the last 8 hours before the procedure,
* Having another chronic disease,
* One-time blood sampling is not performed,
* Fractures or signs of inflammation at acupressure application points

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2022-06-04 (Actual); Primary Completion 2022-06-04 (Actual); Study Completion 2022-06-04 (Actual)

PRIMARY OUTCOMES:
Pain assessment of the child using the Wong Baker Facial Pain Rating scale | Measurements were taken from the scale just before blood was taken.
  The Wong Baker Facial Pain Rating Scale is rated from 0 to 10 (such as 0-2-4-6-8-10). "0" means no pain, and "10" means the most severe pain. This scale is used to diagnose pain in children ages 3-18.
Wong Baker Faces Pain Rating Scale | Measurements were taken just before blood was drawn and a scale was used immediately after blood was drawn.]
  It is applied by explaining to the child that each face belongs to a person, that there is a happy face that does not have any pain, and a sad face that feels a little or a lot of pain. The child is asked to choose the face that best expresses his or her feelings by giving an explanation for each face ("0": he is very happy because he has no pain, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: MELEK GULGUN ALTINTAS, Phd, Principal Investigator — Mersin University
Locations (1):
- Mersin University, Mersin, Yeni̇şehi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study protocol